CLINICAL TRIAL: NCT05884242
Title: Intervention Specific Appendix to PLATFORMPBNAP1001: Evaluation of The Effect of Adalimumab on Inflammatory Mediators Following a Systemic Endotoxin Challenge
Brief Title: A Study of Adalimumab on Inflammatory Mediators Following a Systemic Endotoxin Challenge
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CR109299; 2022-002896-13 (EudraCT Number); NOPRODPBNAP1001 (Other: Janssen Research & Development, LLC); PLATFORMPBNAP1001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2023-05-22; First posted 2023-06-01 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Healthy
MeSH Terms: interventions — Adalimumab; Lipopolysaccharides

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Active Arm: Adalimumab + Lipopolysaccharide (LPS) Challenge (Experimental): Healthy participants will receive adalimumab subcutaneous (SC) injections via prefilled syringe or prefilled pen on Day 1, followed by the LPS intravenous (IV) injection challenge on Day 6.
  Interventions: Drug: Adalimumab; Drug: Lipopolysaccharide (LPS)
- Control Arm: LPS Challenge (Experimental): Participants will receive LPS IV injection on Day 6. No study interaction will be administered.
  Interventions: Drug: Lipopolysaccharide (LPS)

INTERVENTIONS:
Drug: Adalimumab — Adalimumab will be administered subcutaneously.
  Other Names: Humira
  Arms: Active Arm: Adalimumab + Lipopolysaccharide (LPS) Challenge
Drug: Lipopolysaccharide (LPS) — LPS will be administered intravenously.

SUMMARY:
The purpose of the study is to characterize the inflammatory response to lipopolysaccharide (LPS; molecules that contains fats and carbohydrates) in the presence of a targeted immune pathway modulator.

ELIGIBILITY:
Inclusion Criteria:

* A female participant must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during the study and for a period of 5 months after adalimumab administration
* A female participant must agree not to be pregnant or planning to become pregnant while enrolled in this study or within 5 months after the last dose of adalimumab
* Must agree not to receive any vaccinations (including those authorized for emergency use, for example, Coronavirus disease-19 (COVID-19) within 2 weeks after study intervention administration
* A male participant must agree not to plan to father a child while enrolled in this study or within 90 days after the last dose of study intervention
* Has a negative severe acute respiratory syndrome coronavirus 2 (COVID-19) reverse transcription-polymerase chain reaction test within 72 hours prior to adalimumab administration on Day 1
* Otherwise healthy on the basis of physical examination, medical history, and vital signs, and 12-lead electrocardiogram (ECG) performed at screening. Any abnormalities must be considered not clinically significant or consistent with the underlying illness in the study population, as specified in the applicable intervention specific appendix (ISA), and this determination must be recorded in the participant's source documents and initiated by the investigator
* Otherwise healthy on the basis of clinical laboratory tests performed at screening. If the results of the serum chemistry panel, blood coagulation, hematology, or urinalysis are outside the normal reference ranges, the participant may be included only if the investigator judges the abnormalities or deviations from normal to be not clinically significant or to be appropriate and reasonable for the population under study. This determination must be recorded in the participant's source documents and initiated by the investigator

Exclusion Criteria:

* Has a history of congestive heart failure or chronic obstructive pulmonary disease
* Has a history of central or peripheral nervous system demyelinating disease (for example, multiple sclerosis, optic neuritis, or including Guillain-Barre syndrome, respectively)
* Has surgery planned within 10 weeks after the study intervention administration
* Known allergies, hypersensitivity, or intolerance to adalimumab or its excipients
* Had major illness or surgery, (for example, requiring general anesthesia) within 24 weeks before screening, or will not have fully recovered from illness or surgery, or has surgery planned during the time the participant is expected to participate in the study and up to 10 weeks after administration of the study intervention
* History of liver or renal insufficiency significant cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, psychiatric, or metabolic disturbances, unless consistent with the underlying disease of interest in the study population, if applicable
* History of any type of immunodeficiency or autoimmune disease or disease treatment associated with immune suppression or lymphopenia, unless consistent with the underlying disease of interest in the study population, if applicable. These include but are not limited to bone marrow or organ transplantation, lymphoproliferative disorders, T- or B-cell deficiency syndromes, splenectomy, functional asplenia and chronic granulomatous disease
* Has an active, acute, or chronic infection

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-05-22 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-07 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in C-reactive Protein (CRP) | From baseline up to Day 14
  Change from the baseline in CRP levels will be reported.

SECONDARY OUTCOMES:
Change From Baseline Tumour Necrosis Factor-alpha (TNF-alpha) | From baseline up to Day 14
  Change from baseline in TNF-alpha levels will be reported.
Longitudinal Change From Baseline in Temperature | From baseline up to Day 14
  Longitudinal change from baseline in temperature [skin] will be reported.
Longitudinal Change From Baseline in Heart Rate | From baseline up to Day 14
  Longitudinal change from baseline in heart rate will be reported.
Longitudinal Change From Baseline in Blood Pressure | From baseline up to Day 14
  Longitudinal change from baseline in blood pressure will be reported.
Percentage of Participants with Treatment-emergent Adverse Events (TEAEs) | Up to Day 21 (end of study)
  Percentage of participants with TEAEs through Day 14 will be reported. An adverse event (AE) is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the intervention under study. TEAEs are defined as AEs with onset or worsening on or after date of first dose of study treatment.
Percentage of Participants With Treatment-emergent Serious Adverse Events (SAEs) | Up to Day 21 (end of study)
  Percentage of participants with treatment-emergent SAEs will be reported. A SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability or incapacity; congenital anomaly. Treatment-emergent SAEs are defined as serious events between administration of study drug and after the last dose that were absent before treatment or that worsen relative to pretreatment state.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Clinical Pharmacology Unit, Merksem, Belgium

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency